CLINICAL TRIAL: NCT00325819
Title: A Randomized Placebo-controlled Trial of Acetaminophen for Prevention of Post-vaccination Fever in Infants
Brief Title: Acetaminophen Before Vaccines for Infants Study (AVIS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDC Protocol #4665
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Fever
Keywords: Acetaminophen; Vaccination; Immunization
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetaminophen (Active Comparator): Children were randomized 1:1 to receive up to five doses of acetaminophen (10-15mg per kg) or placebo following routine vaccinations.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Children were randomized 1:1 to receive up to five doses of acetaminophen (10-15mg per kg) or placebo following routine vaccinations.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Acetaminophen — Children were randomized 1:1 to receive up to five doses of acetaminophen (10-15mg per kg) or placebo following routine vaccinations.
  Arms: Acetaminophen
Other: placebo — Children were randomized 1:1 to receive up to five doses of acetaminophen (10-15mg per kg) or placebo following routine vaccinations.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see whether giving acetaminophen (the medicine in Tylenol) for routine infant vaccinations is helpful in preventing fever or other symptoms.

DETAILED DESCRIPTION:
Post-vaccination fever occurs in up to 40% of infants receiving routinely recommended childhood vaccinations. Although serious events are rare, post-vaccination fever causes discomfort for the child, can lead to medical utilization, can rarely result in febrile seizure, and can cause a working parent to miss time from their job to care for a febrile infant who cannot attend day care. The benefits of acetaminophen prophylaxis for infants receiving current vaccinations, in terms of reduction of discomfort for the child, improvement of quality-of-life indicators for the parent, or reduction of medical utilization, have not been measured. This randomized, blinded, placebo-controlled trial will assess the efficacy of prophylaxis with acetaminophen in prevention of fever following routine childhood immunizations.

ELIGIBILITY:
Inclusion Criteria:

1. Child is a current Group Health enrollee.
2. Child will be seen at a Group Health clinic for a Well Child visit that is expected to include 2 or more vaccines after 6 wks and before 10 months of age.

Exclusion Criteria:

1. If child was born at less than 36 weeks of gestation, the child is not eligible until 4 months of age or older.
2. If the child's birth weight was less than 5.5 pounds (2500 grams), the child is not eligible until 4 months of age or older.

Ages: 6 Weeks to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 374 (Actual)
Dates: Start 2006-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Jackson, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Result] Jackson LA, Peterson D, Dunn J, Hambidge SJ, Dunstan M, Starkovich P, Yu O, Benoit J, Dominguez-Islas CP, Carste B, Benson P, Nelson JC. A randomized placebo-controlled trial of acetaminophen for prevention of post-vaccination fever in infants. PLoS One. 2011;6(6):e20102. doi: 10.1371/journal.pone.0020102. Epub 2011 Jun 17. PMID 21698100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment took place between May 2006 and September 2009. Children potentially eligible for study participation were identified from the Group Health data systems and parents were mailed a letter providing information on the study.
Pre-assignment Details: No significant events followed participant enrollment prior to group assignment.
Groups:
- Acetaminophen: Children were randomized 1:1 to receive up to five doses of acetaminophen (10-15mg per kg) or placebo following routine vaccinations. Children were to receive a maximum of five doses of the study medication and all doses were to be administered within 24 hours of vaccination. Parents were encouraged to take the bottle of study medication to the vaccination visit, and to give the first dose at that visit, after the child's weight was assessed and within an hour before or after vaccination. Parents were instructed to give subsequent doses a minimum of four hours apart and to give the last dose of study medication no later than 24 hours after vaccination. Following the first dose, each subsequent dose was to be given no earlier than 4 hours following the previous dose. A maximum of five doses of study medication were to be given; the last dose no later than 24 hours after the study vaccination. Study drug was formulated to provide 160 mg of acetaminophen per 5 cc dose.
- Placebo: Children were randomized 1:1 to receive up to five doses of acetaminophen (10-15mg per kg) or placebo following routine vaccinations. Children were to receive a maximum of five doses of the study medication and all doses were to be administered within 24 hours of vaccination. Parents were encouraged to take the bottle of study medication to the vaccination visit, and to give the first dose at that visit, after the child's weight was assessed and within an hour before or after vaccination. Parents were instructed to give subsequent doses a minimum of four hours apart and to give the last dose of study medication no later than 24 hours after vaccination. Following the first dose, each subsequent dose was to be given no earlier than 4 hours following the previous dose. A maximum of five doses of study medication were to be given; the last dose no later than 24 hours after the study vaccination.
Period: Overall Study
Arm/Group | Acetaminophen | Placebo
Started | 185 | 189
Completed | 176 | 176
Not Completed | 9 | 13
Not completed — Study product lost in mail | 2 | 1
Not completed — Did not take a dose of study product | 4 | 9
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Participants who did not receive acetaminophen or placebo due to postal problems (3), who were not given a first dose of acetaminophen or placebo (13) or who were lost to follow-up due to study diary not being returned (6) were not included in analysis.
Groups:
- Acetaminophen: Subjects who were randomized to receive acetaminophen
- Placebo: Subjects who were randomized to receive placebo
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Placebo | Total
Number analyzed (Participants) | 176 | 176 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 176 | 176 | 352
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 24.8 (4.7) | 24.2 (4.7) | 24.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 95 | 172
  Male | 99 | 81 | 180
Region of Enrollment [Number; unit: participants]
  United States | 176 | 176 | 352

OUTCOME MEASURES:

1. Primary Outcome: Fever >=38C Within 32 Hours of Vaccination.
Description: Fever, defined as rectal temperature >=38C within 32 hours of vaccination.
Time Frame: Fever within 32 hours following vaccination
Population: Temperature values were missing for one subject in the acetaminophen group and two subjects in the placebo group.
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 175 | 174
percentage of participants | 14 [0.41 to 1.01] | 22 [0.41 to 1.01]
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; The study sample size of 1000 children was selected to have 80% power to detect a 30% reduction in risk of the primary outcome of rectal temperature >=38 following vaccination. In 2009, during the enrollment period of our trial, another paper reported the results of a randomized trial of acetaminophen prophylaxis in infants which found significantly lower immune responses to various vaccines in the acetaminophen group. In light of thse findings we elected to stop enrollment in our trial; Test type: Superiority or Other; p = 0.053, unadjusted Poisson regression; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.41 to 1.01]

2. Secondary Outcome: Fever >=39C Within 32 Hours of Vaccination.
Description: Fever, defined as rectal temperature >=39C within 32 hours of vaccination.
Time Frame: Fever within 32 hours following vaccination
Population: Temperature values were missing for one subject in the acetaminophen group and two subjects in the placebo group.
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 175 | 174
percentage of participants | 0 | 2
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.08, Fisher Exact; Risk Ratio (RR) = 0

3. Secondary Outcome: Study Assignment Unblinded
Description: The need for unblinding at any time during the study
Time Frame: At any time during participation in the study
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 176 | 176
percentage of participants | 3 | 9
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.02, unadjusted Poisson regression; Risk Ratio (RR) = 0.31, 95% CI 2-sided [0.12 to 0.84]

4. Secondary Outcome: Medical Utilization
Description: Telephone calls to the consulting nurse or the child's physician that were made due to concerns regarding an acute illness, fever, or possible vaccine reaction and outpatient, urgent care, and emergency room visits that were for evaluation of an acute illness, fever, or a possible vaccine reaction, within 32 hours of vaccination.
Time Frame: Within 32 hours of vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 176 | 176
percentage of participants | 3 | 6
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.14, unadjusted Poisson regression; Risk Ratio (RR) = 0.45, 95% CI 2-sided [0.16 to 1.28]

5. Secondary Outcome: Infant Fussiness
Description: Parents were asked to record level of fussiness (compared with the child's usual) within 32 hours of vaccination, using the categories much less than usual, less than usual, about usual, more than usual, and much more than usual.
Time Frame: Within 32 hours of vaccination
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 176 | 176
percentage of participants
  Infant fussiness - About usual or less than usual | 42 | 38
  Infant fussiness-More than or much more than usual | 58 | 62
  Infant fussiness-Much more than usual | 10 | 24
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.001, unadjusted Poisson regression; Risk Ratio (RR) = 0.40, 95% CI 2-sided [0.25 to 0.70]

6. Secondary Outcome: Parent Time Lost From Sleep
Description: Parents were asked about their sleep on the night following the vaccinations. They were asked to report whether they slept much less than usual, less than usual, about the usual amount, more than usual, or much more than usual on that night.
Time Frame: On the night following vaccinations
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 176 | 176
percentage of participants
  Parent sleep - About usual or more than usual | 73 | 77
  Parent sleep - Less than or much less than usual | 27 | 23
  Parent sleep - Much less than usual | 3 | 5
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.40, unadjusted Poisson regression; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.21 to 1.88]

7. Secondary Outcome: Infant Time Lost From Sleep
Description: Parents were asked about their infant's sleep on the night following the vaccinations. They were asked to report whether their infant slept much less than usual, less than usual, about the usual amount, more than usual, or much more than usual on that night.
Time Frame: On the night following vaccinations
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 176 | 176
percentage of participants
  Infant sleep - About usual or more than usual | 78 | 81
  Infant sleep - Less than or much less than usual | 22 | 19
  Infant sleep - Much less than usual | 2 | 2
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 1.00, unadjusted Poisson regression; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.25 to 3.94]

8. Secondary Outcome: Parent Time Lost From Work
Description: Parents were asked to report whether they were scheduled to work on the day of the vaccination visit (but following that visit) or the next day and, if so, whether they had to miss work to care for their infant because of fever, fussiness, or possible vaccine reaction on those days.
Time Frame: Through the day after vaccination
Population: Refers to the number of participants for whom parents reported that they were scheduled to work on the day of the vaccination visit or the day following the child's vaccination visit.
Measure: Number; unit: percentage of participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 143 | 140
percentage of participants | 4 | 1
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.18, unadjusted Poisson regression; Risk Ratio (RR) = 2.94, 95% CI 2-sided [0.60 to 14.34]

ADVERSE EVENTS:
Arm/Group | Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/176
Other Adverse Events (participants affected / at risk) | 0/176 | 0/176

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No